CLINICAL TRIAL: NCT03463590
Title: Deep Brain Stimulation of the Bilateral Habenula for Treatment-Refractory Obsessive-Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of the Department of Functional Neurosurgery, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Habenula DBS for OCD
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Habenula; Obsessive-Compulsive Disorder; Deep brain stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: All subjects will receive bilateral surgical implantation of DBS system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBS (Experimental): All subjects will undergo bilateral surgical implantation of DBS system to habenula. The DBS system will be active at one week after surgery.
  Interventions: Device: Bilateral surgical implantation of DBS system to habenula

INTERVENTIONS:
Device: Bilateral surgical implantation of DBS system to habenula — The DBS device utilized in the present study may include the Medtronic, PINS and SceneRay DBS device depending on patients' choice.

SUMMARY:
Deep brain stimulation (DBS) offers an effective and safe treatment for patients with debilitating, otherwise treatment-refractory obsessive-compulsive disorder(OCD). Although several target areas for DBS have been used for OCD, such as the ventral capsule/ventral striatum and the subthalamic nucleus, not all patients show a clinical response, varying from 10% to 61.5%. Exploring new DBS targets may be a key approach to improve this situation. The habenula is an evolutionarily conserved structure playing an important role in depression, punishment avoiding, reward, addiction, pain and circadian rhythms. The habenula can be considered a promising target for OCD treatment based on the following hypotheses and clinical observations.

1. The lateral habenula DBS has significant clinical antidepressant effects.
2. The habenula plays an important role in the regulation of dopamine and serotonin systems.
3. Selective serotonin reuptake inhibitors, the first line treatment for OCD, are commonly used to treat clinical depression.
4. The habenula serves as a 'negative reward center' that mediates or moderates stress, negative emotions and thoughts, aversive learning, and goal-directed behavior, which are core clinical symptoms and signs of OCD.
5. In our hospital, DBS of the habenula produced a significant improvement in OCD symptoms in one patient who failed to respond to other treatments, including capsulotomy either alone or in combination combined with cingulumotomy.

These theoretical and clinical considerations indicate that the habenula can be seen as a promising DBS target for OCD treatment. This study is focused on the effectiveness of bilateral DBS of the habenula for patients with treatment-refractory OCD. Furthermore, the study is aimed at exploring the influence of DBS of the habenula on brain activity and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having primary OCD according to DSM-IV criteria using the Structured Clinical Interview for DSM-IV Axis I disorders;
* YBOCSII score ≥31；
* Duration ≥2 years；
* Refractoriness to therapy was defined as no response or insufficient response following at least 2 treatments with adequate trials or intolerance to two or three selective serotonin transporter inhibitors (SSRIs) and clomipramine, augmentation strategies (antipsychotics) and cognitive behavioral therapy.
* Capacity to provide informed consent (understanding of the study purpose and methods.

Exclusion Criteria:

* Except for those with major depressive disorder and mild anxiety disorders, patients with clinically significant comorbid DSM-IV diagnoses (such as schizophrenia, bipolar II disorder, alcohol or substance abuse in the last 6 months, current tic disorder, or body dysmorphic disorder)
* Patients with severe personality disorders, assessed using the Structured Clinical Interview for DSM-IV Axis II disorders.
* Serious and unstable organic diseases (e.g. unstable coronal heart disease);
* Pregnancy and/or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Y-BOCSII Score | Baseline (preoperative),1 month, 3 months,6 months, 9 months
  The score of the scale ranges from 0 to 50
Change in OCI-R Score | Baseline (preoperative),1 month, 3 months,6 months, 9 months
  The score of the scale ranges from 0 to 72

SECONDARY OUTCOMES:
changes in the Hamilton Depression Scale(HAMD-17) | Baseline（preoperative）,1 month, 3 months, 6 months,9 months
  The score of the scale ranges from 0 to 50
changes in the Hamilton Anxiety Scale(HAMA-14) | Baseline（preoperative）,1 month, 3 months, 6 months,9 months
  The score of the scale ranges from 0 to 56
changes in FMRI signal | Baseline（preoperative）,3 month, 6 months, 9 months
  The FMRI signal is to estimate Blood Oxygenation Level Dependent (BOLD) and connectivity of brain areas
changes in World Health Organization Quality of Life-BREF(WHO-BREF) | Baseline（preoperative）,1 month, 3 months,6 months,9 months
changes the MOS item short from health survey (SF-36) | Baseline（preoperative）,1 month, 3 months,6 months,9 months
Neuropsychological measures(Scores of cogstate battery) | Baseline（preoperative）,1 month, 3months,6months,9months
  Neuropsychological measures contains six tasks which are detection task, identification task, one card learning task, one back task, Groton maze learning task, set-shifting task

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital Functional Neurosurgery, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Alonso P, Cuadras D, Gabriels L, Denys D, Goodman W, Greenberg BD, Jimenez-Ponce F, Kuhn J, Lenartz D, Mallet L, Nuttin B, Real E, Segalas C, Schuurman R, du Montcel ST, Menchon JM. Deep Brain Stimulation for Obsessive-Compulsive Disorder: A Meta-Analysis of Treatment Outcome and Predictors of Response. PLoS One. 2015 Jul 24;10(7):e0133591. doi: 10.1371/journal.pone.0133591. eCollection 2015. PMID 26208305
- [Background] Kohl S, Baldermann JC. Progress and challenges in deep brain stimulation for obsessive-compulsive disorder. Pharmacol Ther. 2018 Jun;186:168-175. doi: 10.1016/j.pharmthera.2018.01.011. Epub 2018 Jan 31. PMID 29406245
- [Background] Hirschtritt ME, Bloch MH, Mathews CA. Obsessive-Compulsive Disorder: Advances in Diagnosis and Treatment. JAMA. 2017 Apr 4;317(13):1358-1367. doi: 10.1001/jama.2017.2200. PMID 28384832
- [Background] Batalla A, Homberg JR, Lipina TV, Sescousse G, Luijten M, Ivanova SA, Schellekens AFA, Loonen AJM. The role of the habenula in the transition from reward to misery in substance use and mood disorders. Neurosci Biobehav Rev. 2017 Sep;80:276-285. doi: 10.1016/j.neubiorev.2017.03.019. Epub 2017 May 30. PMID 28576510
- [Background] Fakhoury M. The habenula in psychiatric disorders: More than three decades of translational investigation. Neurosci Biobehav Rev. 2017 Dec;83:721-735. doi: 10.1016/j.neubiorev.2017.02.010. Epub 2017 Feb 13. PMID 28223096
- [Background] Antolin-Fontes B, Ables JL, Gorlich A, Ibanez-Tallon I. The habenulo-interpeduncular pathway in nicotine aversion and withdrawal. Neuropharmacology. 2015 Sep;96(Pt B):213-22. doi: 10.1016/j.neuropharm.2014.11.019. Epub 2014 Dec 2. PMID 25476971
- [Background] Boulos LJ, Darcq E, Kieffer BL. Translating the Habenula-From Rodents to Humans. Biol Psychiatry. 2017 Feb 15;81(4):296-305. doi: 10.1016/j.biopsych.2016.06.003. Epub 2016 Jun 7. PMID 27527822